CLINICAL TRIAL: NCT02376712
Title: Diagnostic Value of Urinary Indices in Differentiating Pre-renal and Renal Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bin Du, Director of Medical ICU, Peking Union Medical College Hospital
Other Study IDs: MICU2015-2
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Differential diagnosis; Urinary indices; Renal Blood Flow; Transesophageal Echocardiography
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pre-renal AKI: Three definitions of pre-renal AKI will be used separately:
  1. Hemodynamic instability (any sign of tissue hypoperfusion) on AKI identification, and AKI recovery in 24-72 hours following hemodynamic stabilization.
  2. AKI recovery in less than 72 hours after AKI identification.
  3. Decreased renal blood flow measured by transesophageal echocardiography (TEE).
- Renal AKI: Three definitions of renal AKI will be used separately:
  1. Hemodynamically stable at AKI identification; or hemodynamically instability (any sign of tissue hypoperfusion) on AKI identification, and AKI persistence in 24-72 hours following hemodynamic stabilization.
  2. AKI persistence 72 hours after AKI identification.
  3. Normal or increased renal blood flow measured by TEE.

SUMMARY:
The study aims to evaluate the diagnostic value of urinary indices in differentiating pre-renal and renal acute kidney injury among critically ill patients.

DETAILED DESCRIPTION:
Critically ill patients with acute kidney injury (AKI) will be included. Urinary indices will be obtained immediately after defining AKI, including specific gravity (SG), urine osmolarity (Uosm), urine sodium (UNa), fractional excretion of sodium (FENa), and fractional excretion of urea (FEurea).

The patterns of renal function and hemodynamic status serve as the clinical definition of pre-renal and renal AKI. Hemodynamic status will be evaluated at inclusion and followed during patients' ICU stay. Those who are hemodynamically stable at inclusion are classified as renal AKI. Those who are hemodynamically unstable at inclusion are followed until hemodynamic stabilization. Those with AKI recovery after hemodynamic stabilization are classified as pre-renal AKI. Those without AKI recovery are defined as renal AKI.

Urinary indices are measured again after hemodynamic stability. One of the investigators objectives is to evaluate the diagnostic value of urinary indices using recovery of renal function after hemodynamic stabilization as the definition of pre-renal AKI.

Transesophageal echocardiography (TEE) has been proved to be a reliable method of measuring left renal blood flow during surgical operation. Decreased renal blood flow measured by TEE may serve as an objective definition of pre-renal AKI. The mesurement will be conducted at inclusion if the patient is sedated, intubated, and without TEE contraindication. If the patient is hemodynamically unstable at inclusion, the measurement will be repeated after hemodynamic stabilization. The investigators study also serves the following aims: (1) feasibility of measuring renal blood flow by TEE among critically ill patients; (2) the correspondence between renal blood flow measured by TEE and clinical definition of pre-renal and renal AKI; (3) the diagnostic value of urinary indices in differentiating pre-renal and renal AKI, which is judged by renal blood flow measured by TEE.

ELIGIBILITY:
Inclusion Criteria:

All patients admitted to Medical ICU of PUMCH with one of the following:

* Increase in serum creatinine by ≥ 26.5 umol/l within 48 hours;
* Increase in serum creatinine to ≥ 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days;
* Urine volume < 0.5ml/kg/h for 1 hour.

Exclusion Criteria:

* Obstructive renal disease
* Renal replacement therapy (RRT) for chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed acute kidney injury at ICU admission or during ICU stay
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value of urinary indices in differentiating pre-renal and renal AKI | At ICU admission and during ICU stay
  Urinary indices will be compared between patient groups (pre-renal and renal AKI). Sensitivity analysis will be applied to the cut off values of renal blood flow measured by TEE. Sensitivity and specificity of the indices will be calculated. Receiver operating characteristic curves will be plotted.

SECONDARY OUTCOMES:
Feasibility of measuring renal blood flow among critically ill patients | At ICU admission and during ICU stay
  Feasibility includes rate of success of measurement, intra-observer variability, inter-observer variability, and intraclass correlation coefficients.

OTHER OUTCOMES:
Diagnostic value of urinary indices in the subgroup of patients without diuretic use | At ICU admission and during ICU stay
  The same strategy as the primary outcome will be used in subgroup of patients without diuretic use.
Diagnostic value of urinary indices in the subgroup of patients without sepsis | At ICU admission and during ICU stay
  The same strategy as the primary outcome will be used in subgroup of patients without sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Du, Dr, Principal Investigator — MICU of Peking Union Medical College
Locations (1):
- MICU of Peking Union Medical College, Beijing, China